CLINICAL TRIAL: NCT03426410
Title: Concordance Between the National Recommendations and the Actual Rehabilitation Provided for Low Back Pain Patients Referred to Primary Care Rehabilitation. A Survey of Public and Private Health Care Providers in Denmark
Brief Title: National Recommendations and the Actual Rehabilitation Provided for Low Back Pain Patients
Status: Completed | Type: Observational
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 6500010
Record Dates: First submitted 2018-02-01; First posted 2018-02-08 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-02

CONDITIONS: Guideline Adherence; Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Electronic survey containing a questionnaire regarding knowledge and use of national guidelines of low back pain rehabilitation, type and frequency of cross sectional communication, attitudes and beliefs about back pain and two patient vignettes.

SUMMARY:
Purpose and background:

The purpose of the study is to investigate physiotherapeutic courses of rehabilitation in the primary sector for low back pain patients. This is done by identifying both how physiotherapeutic rehabilitation is organized in the primary sector and further what different types of physiotherapeutic interventions are offered for this patient group. Furthermore the study aims to evaluate to what extent existing physiotherapeutic rehabilitation practice adheres with the national and international guidelines and recommendations for low back pain rehabilitation.

Methods:

A quantitative survey is carried out, which includes development and validation of a questionnaire for the purpose, and this is subsequently distributed electronically to private and public providers of physiotherapy rehabilitation in all 19 municipalities in Central Denmark Region. Approximately 500 physiotherapists will be asked to participate in the survey in the period February to March 2018.

ELIGIBILITY:
Inclusion Criteria:

* physical therapists working with low back pain rehabilitation in the primary sector in Central Denmark Region

Exclusion Criteria:

* physical therapists that have less than 1 consultation per week with low back pain patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study includes physical therapists in Central Denmark Region working with low back pain rehabilitation in the primary sector, either as a public or a private provider.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Guideline adherence | 1 month
  Adherence to guidelines is assessed on the basis of the responses given to the two patient vignettes in the questionnaire. Thus, for each vignette there is a total 3 questions with four possible answers for each question. For each question 1 answer is correct, 1 partly correct and 2 are wrong. Adherence to guidelines is ultimately defined as:
  Strictly adheres = 3 correct answers OR 2 correct and 1 partly correct answer. Partly adheres: 1 correct and 2 partly correct answers OR 2 correct and 1 wrong answer OR 3 partly correct answers.
  Does not adhere: any other combination of answers than the above mentioned.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, PhD, Principal Investigator — Silkeborg Regional Hospital
Locations (1):
- Silkeborg Regional Hospital, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided